CLINICAL TRIAL: NCT06410183
Title: Inter-rater Reliability of Preoperative Mortality Risk Calculators Used for High-risk Noncardiac Surgical Patients
Brief Title: Inter-rater Reliability of Preoperative Mortality Risk Calculators
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Utrecht University (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-2161
Record Dates: First submitted 2024-04-25; First posted 2024-05-13 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Reliability
Keywords: preoperative; high-risk patient

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The goal of this study is to investigate the inter-rater variability of mortality risk calculations for high-risk non-cardiac surgical patients. For this purpose patient information from health care files were used. Five anesthesiologists calculated the mortality risks with three calculators for 34 high-risk non-cardiac surgical patients. The patients were discussed in a preoperative multidisciplinary discussion in a large teaching hospital in The Netherlands.

DETAILED DESCRIPTION:
Identifying high-risk patients for perioperative treatment and decision-making remains a challenge due to difficulty in reliably estimating morbidity and mortality risks. Assessing surgical risk helps allocating resources, obtaining informed consent, and making shared decisions with a multidisciplinary team (MDT). Multimorbidity is increasing globally in an ageing population with a growing burden of chronic diseases. It has been shown that high-risk non-cardiac surgical patients suffer disproportionally from perioperative complications. Preoperative mortality risk calculators are available and may help to identify high-risk non-cardiac surgical patients already before surgery, triggering efforts to lower the burden of possible complications, e.g., by extended monitoring or specified treatments. A systematic review suggested a significant risk of bias in developing current preoperative risk calculators due to lack of external validation, highlighting the need for enhanced performance and reliability to ensure their effectiveness in clinical practice. Low reliability and performance may, despite their general availability, be why that preoperative risk calculators are not yet consistently used in clinical practice. For daily clinical use, good predictive performance, low inter rater variability and user friendliness are essential. Discrepancies in predictor measurements can cause miscalibration, changes in discriminatory ability, and overall accuracy, leading to clinically relevant variability in risk calculator results. Previous studies have shown that physicians must trust a mortality risk calculator before utilization. High-risk patients suffer especially from complications, and it has been shown that the complications often result in death perioperatively. Therefore, adequate preoperative calculation of mortality risks and early recognition of high-risk non-cardiac surgical patients could benefit from reliable preoperative risk calculation. These high-risk patients can then be discussed in a preoperative multidisciplinary discussion to lower complications and perioperative deaths.

The current study evaluated the inter-rater reliability of calculating preoperative mortality risk scores for high-risk non-cardiac surgical patients in clinical practice among five anesthesiologists. The hypothesis was that the available risk calculators would show moderate to good reliability. For this purpose, five anesthesiologists used the following three risk calculators: the preoperative score to predict postoperative morbidity [POSPOM, the American College of Surgeons surgical risk calculator, and the surgical outcome risk tool [SORT].

ELIGIBILITY:
Inclusion Criteria:

* Patients discussed in a preoperative multidisciplinary team (MDT) meeting.

Exclusion Criteria:

* No complete patient file to calculate the mortality risks

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HIgh-risk non-cardiac surgical patients discussed in an MDT meeting.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
inter-rater reliability of three risk calculators: POSPOM, SRC and SORT | After calculation of the mortality risks (1 month)
  Five anesthesiologists calculated mortality risks retrospectively for 34 patients. The intra-class correlation coefficient (ICC) was calculated per risk calculator

SECONDARY OUTCOMES:
mortality risk calculations or 34 patients | 1 month
  the Preoperative scale of postoperative outcome: (POSPOM), the surgical risk calculator: (SRC) and the surgical outcome risk tool: (SORT) mortality risk calculators were used for (retrospective) 30-day mortality risk calculation of 34 patients

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline E. Vernooij, MD, MA, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided